CLINICAL TRIAL: NCT07320443
Title: Platelet Indices in Inflammatory Bowel Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sahar Atef Ahmed Ali, Dr., Assiut University
Other Study IDs: platelet indices in IBD
Record Dates: First submitted 2025-12-04; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic, immune-mediated condition characterized by relapsing inflammation of the gastrointestinal tract. It primarily includes two subtypes: ulcerative colitis (UC) and Crohn's disease (CD), both of which have shown a rising incidence globally over recent decades .The pathogenesis of IBD is complex and multifactorial, involving a dynamic interplay of genetic susceptibility, immune dysregulation, environmental exposures, and gut microbiota alterations .

Recent studies have highlighted the emerging role of platelets beyond hemostasis, particularly in immune modulation and inflammation . Patients with IBD exhibit several platelet-related abnormalities, including changes in platelet count, size, shape, and activation status . These alterations may result from the chronic systemic inflammation characterizing IBD, leading to enhanced platelet reactivity and a prothrombotic state .

Evidence suggests that inflammatory cytokines can trigger coagulation pathways, which in turn amplify inflammation, forming a self-perpetuating cycle . This interplay between inflammation and thrombosis has clinical implications, as IBD patients are at increased risk for thromboembolic events . Mean platelet volume (MPV), plateletcrit (PCT), platelet distribution width (PDW), and platelet count (PLT) are readily accessible indices from a complete blood count that may reflect platelet activity and inflammatory status .

Despite these associations, results from previous studies on platelet indices in IBD patients remain inconsistent. A recent systematic review and meta-analysis demonstrated that MPV is significantly lower in IBD patients compared to healthy controls, while PLT and PCT tend to be elevated .However, the diagnostic and prognostic utility of these indices in clinical practice remains undefined.

DETAILED DESCRIPTION:
we aim to investigate the relationship between platelet indices (MPV, PDW, PCT, PLT) and disease activity in patients with inflammatory bowel disease. We also aim to evaluate the potential correlation between these platelet parameters and established inflammatory markers such as CRP, ESR, and fecal calprotectin. This may help clarify whether platelet indices can serve as accessible, cost-effective biomarkers in the clinical assessment of IBD

ELIGIBILITY:
Inclusion Criteria:

* a. Inclusion criteria:

  * Adult patients (age >18) with confirmed diagnosis of UC , Crohn's b. Exclusion criteria:
* Hematologic malignancies or disorders.
* Pregnancy
* Use of antiplatelet or anticoagulant drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: : Assiut University hospitals IBD out patient clinic and internal medicine department
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
This study aims to evaluate the correlation between platelet indices and disease activity in IBD | From study enrollment up to 5 years.
  Correlation between platelet indices and disease activity in inflammatory bowel disease This study aims to assess the correlation between platelet indices and disease activity in patients with inflammatory bowel disease.
  Platelet indices, including mean platelet volume (MPV), platelet distribution width (PDW), plateletcrit (PCT), and platelet count (PLT), will be measured as continuous variables obtained from complete blood count analysis. Disease activity will be assessed using validated clinical disease activity indices: the Partial Mayo Score for ulcerative colitis and the Crohn's Disease Activity Index (CDAI) for Crohn's disease.
  The correlation between platelet indices and disease activity scores will be evaluated using correlation coefficients (Pearson or Spearman)

SECONDARY OUTCOMES:
Correlation between platelet indices and inflammatory markers in inflammatory bowel disease | From study enrollment up to 5 years
  This study aims to assess the correlation between platelet indices and inflammatory markers in patients with inflammatory bowel disease.
  Platelet indices (MPV, PDW, PCT, and PLT) will be correlated with inflammatory markers, including C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR), using correlation coefficients (Pearson or Spearman).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/39044827/